CLINICAL TRIAL: NCT04567056
Title: Validation of Specific Methylation Profiles Ind Head and Neck Cancer - a Cohort Study
Brief Title: Specific Methylation Profiles in HNSCC
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Christian Sander Danstrup, Associate Professor, M.D., Aalborg University Hospital
Other Study IDs: N-20190047-2
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; Squamous Cell carcinoma; Methylation; DNA
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cancer group: Patients with verified head and neck squamous cell carcinomas
  Interventions: Diagnostic Test: Blood sample
- Control group: Matched control group without active or earlier cancer and a normal ENT examination.
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — A separate blood sample will be taken for methylation-analyses

SUMMARY:
In the study, N-20190047, the investigators aim to define specific methylation patterns in a group of patients with head and neck squamous cell carcinomas.

With this study the investigators aim to validate these findings in a larger cohort.

ELIGIBILITY:
Cancer group:

Inclusion Criteria:

* Written informed consent
* Verified head and neck squamous cell carcinoma

Exclusion Criteria:

* Other active cancer
* Uncontrolled comorbidity
* Unable to give informed consent

Control group:

Inclusion Criteria:

* Written informed consent
* Normal ENT-examination

Exclusion Criteria:

* Other active cancer
* Uncontrolled comorbidity
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer group:
  Patients referred from the region of Northern Denmark to the Department of Otorhinolaryngology - Head and Neck Surgery with suspicion of, or with already verified Head and neck squamous cell carcinoma. Only patients with verified squamous cell carcinoma after diagnostic work-up will be eligible.
  Control group:
  Patients referred from the region of Northern Denmark to the Department of Otorhinolaryngology - Head and Neck Surgery for evaluation or treatment, but without suspected or verified malignancy of the head and neck.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | At diagnosis
  How accurate can the methylation profiles diagnose the head and neck squamous cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gaihede, Professor, Principal Investigator — Department of Otolaryngology - Head and Neck Surgery, Aalborg University Hospital
Locations (1):
- Department of Otolaryngology - Head and Neck Surgery, Aalborg, Denmark